CLINICAL TRIAL: NCT01431313
Title: A Dose Escalation Study to Evaluate the Effect of Inhaled Nitrite on Cardiopulmonary Hemodynamics in Subjects With Pulmonary Hypertension
Brief Title: Inhaled Nitrite in Subjects With Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Schmidhofer, Mark, MD (Individual)
Responsible Party: Principal Investigator, Marc A. Simon, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO11080686
Record Dates: First submitted 2011-09-06; First posted 2011-09-09 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Hypertension; Heart Failure, Diastolic
Keywords: pulmonary hypertension; heart failure
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure, Diastolic; Heart Failure | interventions — Sodium Nitrite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inhaled Nitrite (Experimental): Sodium Nitrite Inhalation Solution (AIR001) 45mg dosage with one subsequent escalation dosage of 90mg based on tolerability.
  Interventions: Drug: Inhaled Nitrite

INTERVENTIONS:
Drug: Inhaled Nitrite — Each patient will receive a starting dose of 45 mg of inhaled nitrite, with one planned subsequent planned dose of 90 mg of inhaled nitrite
  Other Names: Sodium Nitrite

SUMMARY:
This is a single-center, open label phase II study to evaluate the effect of inhaled nitrite delivered in a dose escalation manner on the change in pulmonary vascular resistance (PVR) in subjects with pulmonary hypertension undergoing right heart catheterization.

A total of 50 subjects with a confirmed diagnosis of pulmonary hypertension and meet all inclusion/exclusion criteria will be enrolled in the study which will entail a single right heart catheterization and nebulized nitrite dose of 45mg with one subsequent dosage of 90 mg.

DETAILED DESCRIPTION:
Screening Visit:Initial screening evaluations including physical examination, medical history, and clinical laboratory assessments will be conducted to determine study eligibilities during a routine clinic visit at the UPMC HVI, CLC or inpatient at UPMC Presbyterian. Subjects who meet the inclusion criteria and none of the exclusion criteria will be entered into the study.

Day 1: This study visit will occur on the same day subjects are scheduled for their clinically indicated right heart catheterization or who volunteer for a research right heart catheterization for this specific study. Subjects on oral background PAH therapy (ETRA or PDE5I) will be instructed to hold their regimen on the day of the study visit.

Subjects will receive nebulized AIR001 doses escalated based upon safety and tolerability. The dose of inhaled nitrite will be delivered via electronic nebulizer. During the study right heart/pulmonary artery hemodynamics will be measured as well as noninvasive systemic blood pressure monitoring. Subjects will be tested for the changes in pulmonary vascular resistance (PVR) using standard clinical protocol hemodynamic recordings of right atrial, right ventricular, and pulmonary artery pressures, in addition to cardiac output at time zero,

3 Day phone follow up

30 Day follow up visit: All subjects enrolled in the study will be followed for 30 days (+/- 5 day window) after completion of the study treatment. A physical exam and clinical labs will be obtained at this visit.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of RHC confirmed WHO Group I PAH n=20

Idiopathic, primary or familial pulmonary arterial hypertension PAH associated with one of the following connective tissue diseases:

PAH associated with exposure to drugs and toxins eg, anorexigens, L-tryptophan, toxic rapeseed oil Stable PAH for at least 3 months if on therapy This patient population is closed to enrollment. Target enrollment of 20 subjects has been met

WHO Group II Pulmonary Hypertension n=20 Pulmonary capillary wedge pressure PWCP greater than 15 AND Transpulmonary Gradient TPG greater than12

WHO Group III PH n = 10

* Has WHO functional class II through IV symptoms
* Had the diagnosis of PH confirmed by a cardiac catheterization Both WHO Group I PAH and WHO Group III PH

WHO GROUP I PAH, II and III PH Age 18 and older Able to participate in right heart catheterization Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria

Age less than 18 years

Baseline systemic hypotension, defined as MAP less than 50 mmHg

Required intravenous inotropes within 30 days prior to study participation;

Has uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure greater than160 mm Hg or sitting diastolic blood pressure greater than100 mm Hg at screening

Has a history of portal hypertension or chronic liver disease, including hepatitis B and/or hepatitis C with evidence of recent infection and/or active virus replication defined as moderate to severe hepatic impairment Child-Pugh Class B-C

Has chronic renal insufficiency as defined by serum creatinine greater than 2.5 mgdL at screening or requires dialytic support

Has a hemoglobin concentration less than 9 gdL at Screening

History of atrial septostomy within 6 months prior to Day 1 visit

Repaired or unrepaired congenital heart disease CHD

Pericardial constriction

Confirmed diagnosis of restrictive or congestive cardiomyopathy;

Left ventricular ejection fraction 40 percent by multiple gated acquisition scan MUGA, angiography or echocardiography

Symptomatic coronary disease with demonstrable ischemia;

Other severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study

Has a psychiatric, addictive or other disorder that compromises the ability to give informed consent for participating in this study. This includes subjects with a recent history of abusing alcohol or illicit drugs 30 days prior to study screening Day 0and for the duration of the study

Poorly controlled asthma defined by active wheezing and or cough with FEV1 less than 70 percent predicted, responsive to inhaled BD greater than 15 percent increase in FEV1 with BD

Investigators, study staff or their immediate families

Clinically significant intercurrent illness (including lower respiratory tract infection) or clinically significant surgery within 4 weeks before the administration of study drug

Personal or family history of congenital or acquired methemoglobinemia

Personal or family history of RBC CYP B5 reductase deficiency

Known or suspected hypersensitivity or allergic reaction to sodium nitrite Personal history of glucose-6-phosphate dehydrogenase G6PD deficiency or any contraindication to receiving methylene blue

If female, is pregnant or breast feeding, or has a positive pregnancy test result predose

Receipt of an investigational product or device, or participation in a drug research study within a period of 15 days or 5 half-lives of the drug, whichever is longer before the first dose of study drug

Blood loss or blood donation greater than 550 mL within 90 days or plasma donation greater than 500 mL within 14 days before administration of study drug

RHC less than 2 weeks from treatment visit unless clinically indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc A. Simon, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] DeMartino AW, Kim-Shapiro DB, Patel RP, Gladwin MT. Nitrite and nitrate chemical biology and signalling. Br J Pharmacol. 2019 Jan;176(2):228-245. doi: 10.1111/bph.14484. Epub 2018 Oct 3. PMID 30152056
- [Background] Gladwin MT. How Red Blood Cells Process Nitric Oxide: Evidence for the Nitrite Hypothesis. Circulation. 2017 Jan 10;135(2):177-179. doi: 10.1161/CIRCULATIONAHA.116.024752. No abstract available. PMID 28069711
- [Background] Lai YC, Tabima DM, Dube JJ, Hughan KS, Vanderpool RR, Goncharov DA, St Croix CM, Garcia-Ocana A, Goncharova EA, Tofovic SP, Mora AL, Gladwin MT. SIRT3-AMP-Activated Protein Kinase Activation by Nitrite and Metformin Improves Hyperglycemia and Normalizes Pulmonary Hypertension Associated With Heart Failure With Preserved Ejection Fraction. Circulation. 2016 Feb 23;133(8):717-31. doi: 10.1161/CIRCULATIONAHA.115.018935. Epub 2016 Jan 26. PMID 26813102
- [Background] Hon YY, Lin EE, Tian X, Yang Y, Sun H, Swenson ER, Taveira-Dasilva AM, Gladwin MT, Machado RF. Increased consumption and vasodilatory effect of nitrite during exercise. Am J Physiol Lung Cell Mol Physiol. 2016 Feb 15;310(4):L354-64. doi: 10.1152/ajplung.00081.2015. Epub 2015 Dec 18. PMID 26684248
- [Background] Vanderpool R, Gladwin MT. Harnessing the nitrate-nitrite-nitric oxide pathway for therapy of heart failure with preserved ejection fraction. Circulation. 2015 Jan 27;131(4):334-6. doi: 10.1161/CIRCULATIONAHA.114.014149. Epub 2014 Dec 22. No abstract available. PMID 25533965
- [Background] Rix PJ, Vick A, Attkins NJ, Barker GE, Bott AW, Alcorn H Jr, Gladwin MT, Shiva S, Bradley S, Hussaini A, Hoye WL, Parsley EL, Masamune H. Pharmacokinetics, pharmacodynamics, safety, and tolerability of nebulized sodium nitrite (AIR001) following repeat-dose inhalation in healthy subjects. Clin Pharmacokinet. 2015 Mar;54(3):261-72. doi: 10.1007/s40262-014-0201-y. PMID 25421879
- [Background] Bueno M, Wang J, Mora AL, Gladwin MT. Nitrite signaling in pulmonary hypertension: mechanisms of bioactivation, signaling, and therapeutics. Antioxid Redox Signal. 2013 May 10;18(14):1797-809. doi: 10.1089/ars.2012.4833. Epub 2012 Oct 15. PMID 22871207
- [Background] Totzeck M, Hendgen-Cotta UB, Luedike P, Berenbrink M, Klare JP, Steinhoff HJ, Semmler D, Shiva S, Williams D, Kipar A, Gladwin MT, Schrader J, Kelm M, Cossins AR, Rassaf T. Nitrite regulates hypoxic vasodilation via myoglobin-dependent nitric oxide generation. Circulation. 2012 Jul 17;126(3):325-34. doi: 10.1161/CIRCULATIONAHA.111.087155. Epub 2012 Jun 9. PMID 22685116
- [Background] Sparacino-Watkins CE, Lai YC, Gladwin MT. Nitrate-nitrite-nitric oxide pathway in pulmonary arterial hypertension therapeutics. Circulation. 2012 Jun 12;125(23):2824-6. doi: 10.1161/CIRCULATIONAHA.112.107821. Epub 2012 May 9. No abstract available. PMID 22572912
- [Background] Zuckerbraun BS, George P, Gladwin MT. Nitrite in pulmonary arterial hypertension: therapeutic avenues in the setting of dysregulated arginine/nitric oxide synthase signalling. Cardiovasc Res. 2011 Feb 15;89(3):542-52. doi: 10.1093/cvr/cvq370. Epub 2010 Dec 22. PMID 21177703
- [Background] Lundberg JO, Weitzberg E, Gladwin MT. The nitrate-nitrite-nitric oxide pathway in physiology and therapeutics. Nat Rev Drug Discov. 2008 Feb;7(2):156-67. doi: 10.1038/nrd2466. PMID 18167491
- [Background] Dejam A, Hunter CJ, Tremonti C, Pluta RM, Hon YY, Grimes G, Partovi K, Pelletier MM, Oldfield EH, Cannon RO 3rd, Schechter AN, Gladwin MT. Nitrite infusion in humans and nonhuman primates: endocrine effects, pharmacokinetics, and tolerance formation. Circulation. 2007 Oct 16;116(16):1821-31. doi: 10.1161/CIRCULATIONAHA.107.712133. Epub 2007 Sep 24. PMID 17893272
- [Background] Vangeneugden T, Laenen A, Geys H, Renard D, Molenberghs G. Applying linear mixed models to estimate reliability in clinical trial data with repeated measurements. Control Clin Trials. 2004 Feb;25(1):13-30. doi: 10.1016/j.cct.2003.08.009. PMID 14980746
- [Result] Simon MA, Vanderpool RR, Nouraie M, Bachman TN, White PM, Sugahara M, Gorcsan J 3rd, Parsley EL, Gladwin MT. Acute hemodynamic effects of inhaled sodium nitrite in pulmonary hypertension associated with heart failure with preserved ejection fraction. JCI Insight. 2016 Nov 3;1(18):e89620. doi: 10.1172/jci.insight.89620. PMID 27812547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in the trial between June 2012 and October 2017.
Groups:
- WHO Group I PAH: Idiopathic, primary or familial pulmonary arterial hypertension PAH associated with one of the following connective tissue diseases: PAH associated with exposure to drugs and toxins eg, anorexigens, L-tryptophan, toxic rapeseed oil. Stable PAH for at least 3 months if on therapy. Additionally, the mean pulmonary artery pressure (MPAP) ≥ 25 mm Hg, pulmonary capillary wedge pressure (PCWP) ≤ 15 mm Hg, and pulmonary vascular resistance (PVR) ≥ 3 Woods units.
  Sodium Nitrite Inhalation Solution (AIR001) 45mg dosage with one subsequent escalation dosage of 90mg based on tolerability.
- WHO Group II Pulmonary Hypertension (PH): MPAP ≥ 25 mm Hg, PWCP > 15, and Transpulmonary Gradient (TPG) > 12. Additionally, LVEF ≥ 40% and dyspnea resulting at least a mild limitation to physical activity (functional class II or greater).
  Sodium Nitrite Inhalation Solution (AIR001) 45mg dosage with one subsequent escalation dosage of 90mg based on tolerability.
- WHO Group III PH: MPAP ≥ 25 mm Hg, PCWP ≤ 15 mm Hg, and PVR ≥ 3 Woods units.
  Sodium Nitrite Inhalation Solution (AIR001) 45mg dosage with one subsequent escalation dosage of 90mg based on tolerability.
Period: Overall Study
Arm/Group | WHO Group I PAH | WHO Group II Pulmonary Hypertension (PH) | WHO Group III PH
Started | 20 | 20 | 8
Completed | 20 | 20 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- WHO Group II PH: MPAP ≥ 25 mm Hg, PWCP > 15, and Transpulmonary Gradient (TPG) > 12. Additionally, LVEF ≥ 40% and dyspnea resulting at least a mild limitation to physical activity (functional class II or greater).
  Sodium Nitrite Inhalation Solution (AIR001) 45mg dosage with one subsequent escalation dosage of 90mg based on tolerability.
- Total: Total of all reporting groups
Arm/Group | WHO Group I PAH | WHO Group II PH | WHO Group III PH | Total
Number analyzed (Participants) | 20 | 20 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (13) | 70 (7) | 68 (6) | 64 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 3 | 25
  Male | 7 | 11 | 5 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 7 | 47
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 19 | 20 | 6 | 45
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Vascular Resistance (PVR)
Description: Linear mixed effects model across all time points and doses relative to baseline. The mixed effects model takes into account all time points combined (repeated measures) and has been extensively described for clinical trials (please see references). In this model, the effect of treatment on hemodynamics (measured at 0, 15, 30, 45, and 60 minutes after 45mg followed by same times after 90 mg dose) was compared with baseline values. We assessed the overall linear trend of treatment. The effect of treatment on hemodynamics in each patient group was assessed separately in mixed-effects models. Since pulmonary vascular resistance (PVR) was not normally distributed, it was transformed to natural log prior to analysis. The reported mean is the change from baseline of PVR over all subsequent times and doses (beta from the mixed effects model, converted back from natural log to Woods units), and is reported as the mean and 95% confidence interval.
Time Frame: Time zero, 15, 30, 45 and 60 minutes after nebulization of 45mg followed by 90 mg dose
Measure: Mean (95% Confidence Interval); unit: Woods units
Groups:
- WHO Group I Pulmonary Arterial Hypertension (PAH): Idiopathic, primary or familial pulmonary arterial hypertension (PAH) associated with one of the following connective tissue diseases: PAH associated with exposure to drugs and toxins eg, anorexigens, L-tryptophan, toxic rapeseed oil. Stable PAH for at least 3 months if on therapy. Additionally, the mean pulmonary artery pressure (MPAP) ≥ 25 mm Hg, pulmonary capillary wedge pressure (PCWP) ≤ 15 mm Hg, and pulmonary vascular resistance (PVR) ≥ 3 Woods units.
  Sodium Nitrite Inhalation Solution (AIR001) 45mg dosage with one subsequent escalation dosage of 90mg based on tolerability.
- WHO Group II Pulmonary Hypertension (PH): mean pulmonary artery pressure (MPAP) ≥ 25 mm Hg, pulmonary capillary wedge pressure (PCWP) > 15, and Transpulmonary Gradient (TPG) > 12. Additionally, left ventricular ejection fraction (LVEF) ≥ 40% and dyspnea resulting at least a mild limitation to physical activity (functional class II or greater).
  Sodium Nitrite Inhalation Solution (AIR001) 45mg dosage with one subsequent escalation dosage of 90mg based on tolerability.
- WHO Group III Pulmonary Hypertension (PH): mean pulmonary artery pressure (MPAP) ≥ 25 mm Hg, pulmonary capillary wedge pressure (PCWP) ≤ 15 mm Hg, and pulmonary vascular resistance (PVR) ≥ 3 Woods units.
  Sodium Nitrite Inhalation Solution (AIR001) 45mg dosage with one subsequent escalation dosage of 90mg based on tolerability.
Arm/Group | WHO Group I Pulmonary Arterial Hypertension (PAH) | WHO Group II Pulmonary Hypertension (PH) | WHO Group III Pulmonary Hypertension (PH)
Number analyzed (Participants) | 20 | 20 | 8
Woods units | 0.77 [0.28 to 1.26] | 0.40 [0.07 to 0.74] | -0.39 [-0.93 to 0.16]
Statistical Analysis 1: Comparison: WHO Group I Pulmonary Arterial Hypertension (PAH); Test type: Other — Mixed effects model across all time points; p = 0.002, Mixed Models Analysis
Statistical Analysis 2: Comparison: WHO Group II Pulmonary Hypertension (PH); Test type: Other — Mixed effects model across all time points; p = 0.003, Mixed Models Analysis
Statistical Analysis 3: Comparison: WHO Group III Pulmonary Hypertension (PH); Test type: Other — Mixed effects model across all time points; p = 0.66, Mixed Models Analysis

2. Secondary Outcome: Time to Maximum Pulmonary Vascular Resistance (PVR) Decrease
Description: Time in minutes to maximum PVR decrease. During study procedure, hemodynamics were measured at 0, 15, 30, 45, and 60 minutes after 45 mg followed by same times after 90 mg dose. The time point at which each patient's maximal decrease in PVR occurred was recorded and reported as the mean and standard deviation in each cohort.
Time Frame: 0, 15, 30, 45, and 60 minutes after 45 mg followed by same times after 90 mg dose
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- WHO Group I Pulmonary Arterial Hypertension (PAH): Idiopathic, primary or familial pulmonary arterial hypertension PAH associated with one of the following connective tissue diseases: PAH associated with exposure to drugs and toxins eg, anorexigens, L-tryptophan, toxic rapeseed oil. Stable PAH for at least 3 months if on therapy. Additionally, the mean pulmonary artery pressure (MPAP) ≥ 25 mm Hg, pulmonary capillary wedge pressure (PCWP) ≤ 15 mm Hg, and pulmonary vascular resistance (PVR) ≥ 3 Woods units.
  Sodium Nitrite Inhalation Solution (AIR001) 45mg dosage with one subsequent escalation dosage of 90mg based on tolerability.
Arm/Group | WHO Group I Pulmonary Arterial Hypertension (PAH) | WHO Group II Pulmonary Hypertension (PH) | WHO Group III Pulmonary Hypertension (PH)
Number analyzed (Participants) | 20 | 20 | 8
minutes | 42.0 (19.2) | 33.0 (17.9) | 42.5 (14.1)

3. Secondary Outcome: Change in Systemic Blood Pressure (Mean Arterial Pressure, MAP)
Description: Linear mixed effects model across all time points and doses relative to baseline. The mixed effects model takes into account all time points combined (repeated measures) and has been extensively described for clinical trials (please see references). In this model, the effect of treatment on hemodynamics (measured at 0, 15, 30, 45, and 60 minutes after 45mg followed by same times after 90 mg dose) was compared with baseline values. We assessed the overall linear trend of treatment. The effect of treatment on hemodynamics in each patient group was assessed separately in mixed-effects models. The reported mean is the change from baseline of MAP over all subsequent times and doses (beta from the mixed effects model), and is reported as the mean and 95% confidence interval.
Time Frame: Time zero, 15, 30, 45 and 60 minutes after nebulization of 45mg followed by 90 mg dose
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | WHO Group I Pulmonary Arterial Hypertension (PAH) | WHO Group II Pulmonary Hypertension (PH) | WHO Group III Pulmonary Hypertension (PH)
Number analyzed (Participants) | 20 | 20 | 8
mmHg | -5.1 [-7.6 to -2.6] | -3.4 [-6.6 to -0.3] | -9.5 [-13.1 to -6.0]
Statistical Analysis 1: Comparison: WHO Group I Pulmonary Arterial Hypertension (PAH); Test type: Other — Mixed effects model across all time points; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: WHO Group II Pulmonary Hypertension (PH); Test type: Other — Mixed effects model across all time points; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: WHO Group III Pulmonary Hypertension (PH); Test type: Other — Mixed effects model across all time points; p < 0.001, Mixed Models Analysis

4. Secondary Outcome: Change in Systemic Vascular Resistance (SVR)
Description: Linear mixed effects model across all time points and doses relative to baseline. The mixed effects model takes into account all time points combined (repeated measures) and has been extensively described for clinical trials (please see references). In this model, the effect of treatment on hemodynamics (measured at 0, 15, 30, 45, and 60 minutes after 45mg followed by same times after 90 mg dose) was compared with baseline values. We assessed the overall linear trend of treatment. The effect of treatment on hemodynamics in each patient group was assessed separately in mixed-effects models. Since systemic vascular resistance was not normally distributed, it was transformed to natural log prior to analysis. The reported mean is the change from baseline of SVR over all subsequent times and doses (beta from the mixed effects model), and is reported as the mean and 95% confidence interval.
Time Frame: Time zero, 15, 30, 45 and 60 minutes after nebulization of 45mg followed by 90 mg dose
Measure: Mean (95% Confidence Interval); unit: mmHg⋅min/L
Arm/Group | WHO Group I Pulmonary Arterial Hypertension (PAH) | WHO Group II Pulmonary Hypertension (PH) | WHO Group III Pulmonary Hypertension (PH)
Number analyzed (Participants) | 20 | 20 | 8
mmHg⋅min/L | -0.43 [-1.42 to 0.55] | 1.19 [0.21 to 2.15] | -2.04 [-3.40 to -0.67]
Statistical Analysis 1: Comparison: WHO Group I Pulmonary Arterial Hypertension (PAH); Test type: Other — Mixed effects model across all time points; p = 0.8, Mixed Models Analysis
Statistical Analysis 2: Comparison: WHO Group II Pulmonary Hypertension (PH); Test type: Other — Mixed effects model across all time points; p = 0.01, Mixed Models Analysis
Statistical Analysis 3: Comparison: WHO Group III Pulmonary Hypertension (PH); Test type: Other — Mixed effects model across all time points; p = 0.01, Mixed Models Analysis

5. Secondary Outcome: Change in Pulmonary Vascular Impedance / Wave Intensity
Description: Characteristic impedance (Zc) which may be related to compliance effects in the large, conduit arteries.
Time Frame: Pre dose and 60 minutes post last dosage inhaled
Population: Data are reported in each group for the subset in whom this data was collected.
Measure: Median (95% Confidence Interval); unit: dyne*sec/cm5
Arm/Group | WHO Group I Pulmonary Arterial Hypertension (PAH) | WHO Group II Pulmonary Hypertension (PH) | WHO Group III Pulmonary Hypertension (PH)
Number analyzed (Participants) | 20 | 14 | 6
dyne*sec/cm5 | -0.004 [-1.02 to 0.33] | -0.34 [-0.83 to -0.02] | -0.20 [-0.69 to 0.29]
Statistical Analysis 1: Comparison: WHO Group I Pulmonary Arterial Hypertension (PAH); Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: WHO Group II Pulmonary Hypertension (PH); Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: WHO Group III Pulmonary Hypertension (PH); Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Plasma Nitrite Concentrations in Mixed Venous Blood
Description: Linear mixed effects model across all time points and doses relative to baseline. The mixed effects model takes into account all time points combined (repeated measures) and has been extensively described for clinical trials (please see references). In this model, the effect of treatment on hemodynamics (measured at 0, 15, 30, 45, and 60 minutes after 45mg followed by same times after 90 mg dose) was compared with baseline values. We assessed the overall linear trend of treatment. The effect of treatment on hemodynamics in each patient group was assessed separately in mixed-effects models. The reported mean is the change from baseline of plasma nitrite concentrations in mixed venous blood over all subsequent times and doses (beta from the mixed effects model), and is reported as the mean and 95% confidence interval.
Time Frame: Pre-dose, 15 minutes post 45mg and 90mg inhalation
Population: Data are reported in each group for the subset in whom this data was collected.
Measure: Mean (95% Confidence Interval); unit: micromolar
Arm/Group | WHO Group I Pulmonary Arterial Hypertension (PAH) | WHO Group II Pulmonary Hypertension (PH) | WHO Group III Pulmonary Hypertension (PH)
Number analyzed (Participants) | 18 | 20 | 6
micromolar | 9.9 [7.4 to 12.5] | 7.0 [4.7 to 9.2] | 7.4 [2.7 to 12.1]
Statistical Analysis 1: Comparison: WHO Group I Pulmonary Arterial Hypertension (PAH); Test type: Other — Mixed effects model of concentrations measured at Pre-dose, 15 minutes post 45mg dose and 15 minutes post 90mg dose; p < 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: WHO Group II Pulmonary Hypertension (PH); Test type: Other — Mixed effects model of concentrations measured at Pre-dose, 15 minutes post 45mg dose and 15 minutes post 90mg dose; p < 0.05, Mixed Models Analysis
Statistical Analysis 3: Comparison: WHO Group III Pulmonary Hypertension (PH); Test type: Other — Mixed effects model of concentrations measured at Pre-dose, 15 minutes post 45mg dose and 15 minutes post 90mg dose; p < 0.05, Mixed Models Analysis

7. Secondary Outcome: Change in Pulmonary Artery Occlusion (Capillary) Pullback Nitrite
Description: Linear mixed effects model across all time points and doses relative to baseline. The mixed effects model takes into account all time points combined (repeated measures) and has been extensively described for clinical trials (please see references). In this model, the effect of treatment on hemodynamics (measured at 0, 15, 30, 45, and 60 minutes after 45mg followed by same times after 90 mg dose) was compared with baseline values. We assessed the overall linear trend of treatment. The effect of treatment on hemodynamics in each patient group was assessed separately in mixed-effects models. The reported mean is the change from baseline of pulmonary artery occlusion (capillary) pullback nitrite concentration over all subsequent times and doses (beta from the mixed effects model), and is reported as the mean and 95% confidence interval.
Time Frame: Pre-dose, 15 minutes post 45mg and 90mg inhalation
Population: Data are reported only for WHO Group I PAH and WHO Group III Pulmonary Hypertension (PH), as there was insufficient data for this analysis for WHO Group II PH. Data are reported in each group for the subset in whom this data was collected.
Measure: Mean (95% Confidence Interval); unit: micromolar
Arm/Group | WHO Group I Pulmonary Arterial Hypertension (PAH) | WHO Group II Pulmonary Hypertension (PH) | WHO Group III Pulmonary Hypertension (PH)
Number analyzed (Participants) | 9 | 0 | 3
micromolar | 9.2 [6.2 to 12.1] |  | 2.4 [0.04 to 4.7]
Statistical Analysis 1: Comparison: WHO Group I Pulmonary Arterial Hypertension (PAH); Test type: Other — Mixed effects model of concentrations measured at Pre-dose, 15 minutes post 45mg dose and 15 minutes post 90mg dose; p < 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: WHO Group III Pulmonary Hypertension (PH); Test type: Other — Mixed effects model of concentrations measured at Pre-dose, 15 minutes post 45mg dose and 15 minutes post 90mg dose; p < 0.001, Mixed Models Analysis

8. Secondary Outcome: Change in Mitochondrial Oxygen Consumption Compared to Baseline After Each Dose of Nitrite
Description: Basal platelet oxygen consumption measured in isolated platelets by extracellular flux analysis (XF24, Seahorse Biosciences, Billerica, MA).
Time Frame: Maximal effect at 15 minutes post 45mg or 90mg inhalation vs Pre dose
Population: Data are reported in each group for the subset in whom this data was collected.
Measure: Mean (95% Confidence Interval); unit: picomoles O2/min
Arm/Group | WHO Group I Pulmonary Arterial Hypertension (PAH) | WHO Group II Pulmonary Hypertension (PH) | WHO Group III Pulmonary Hypertension (PH)
Number analyzed (Participants) | 6 | 16 | 1
picomoles O2/min | -17.58 [-29.66 to -5.50] | 8.62 [-4.97 to 22.21] | -11.64 [-54.12 to 30.83]
Statistical Analysis 1: Comparison: WHO Group I Pulmonary Arterial Hypertension (PAH); Test type: Other — Mixed effects model across all doses; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: WHO Group II Pulmonary Hypertension (PH); Test type: Other — Mixed effects model across all doses; p = 0.21, Mixed Models Analysis
Statistical Analysis 3: Comparison: WHO Group III Pulmonary Hypertension (PH); Test type: Other — Mixed effects model across all doses; p = 0.59, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 30 days +/- 5 days from Right Heart Catheterization
Arm/Group | WHO Group I Pulmonary Arterial Hypertension (PAH) | WHO Group II Pulmonary Hypertension (PH) | WHO Group III Pulmonary Hypertension (PH)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/8
Other Adverse Events (participants affected / at risk) | 4/20 | 6/20 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WHO Group I Pulmonary Arterial Hypertension (PAH) (N=20) | WHO Group II Pulmonary Hypertension (PH) (N=20) | WHO Group III Pulmonary Hypertension (PH) (N=8)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Lightheaded/Dizziness (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Back/neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
increase in serum creatinine from baseline (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small, early phase II pilot study, limited number of subjects. Exercise hemodynamics would be helpful in this population. Findings of acute changes in hemodynamics may or may not be translatable to chronic administration and longer-term outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT01431313/Prot_SAP_000.pdf